CLINICAL TRIAL: NCT00740883
Title: Eighteen Months of Oral Anticoagulant Therapy Versus Placebo After 6 Six Months of Anticoagulation for a First Episode of Idiopathic Pulmonary Embolism: a Multicentre Double-blind Randomized Controlled Trial. "PADIS-PE" Study.
Brief Title: Extended Duration of Oral Anticoagulant Therapy After a First Episode of Idiopathic Pulmonary Embolism: a Randomized Controlled Trial. "PADIS-PE" Study.
Acronym: PADIS EP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RB06.076
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Embolism
Keywords: venous thromboembolism; warfarin; duration of anticoagulation; recurrent venous thromboembolism; anticoagulant-related bleeding
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 18 months of active warfarin therapy
  Interventions: Drug: warfarin
- 2 (Placebo Comparator): 18 months of placebo of warfarin
  Interventions: Drug: placebo of warfarin

INTERVENTIONS:
Drug: warfarin — 18 months of warfarin therapy, once daily
  Arms: 1
Drug: placebo of warfarin — 18 months of placebo of warfarin therapy, once daily
  Arms: 2

SUMMARY:
Rational: After 3 or 6 months of oral anticoagulation for an episode of acute venous thromboembolism (VTE), the risk of recurrent VTE is high (10 to 15% per year) in comparison with a low risk of recurrence if VTE was provoked by a major transient risk factor such as recent surgery (3% per year) independently of the initial presentation (deep vein thrombosis or pulmonary embolism). After a first episode of idiopathic VTE, 3 months of anticoagulation is associated with a very high risk of recurrence (27% per year); however, the benefit-risk of extended duration of anticoagulation (1 to 2 years) remains uncertain, mainly in relation with an increased risk of anticoagulant related bleeding. Therefore, the last ACCP conference group recommended 6 months of oral anticoagulant therapy after a first episode of idiopathic VTE. However, this recommendation is likely to be inadequate for at least two main reasons: (1) no studies compared 2 years to 6 months of anticoagulation after idiopathic VTE; and (2), if the frequency of recurrent VTE is similar after deep vein thrombosis and pulmonary embolism, however, the case fatality rate of recurrent VTE is higher after pulmonary embolism (12%) than after deep vein thrombosis (5%).

Objective : the main objective is to demonstrate that, after 6 months of oral anticoagulation for a first episode of idiopathic pulmonary embolism, 18 months of warfarin therapy is associated with a lower cumulative risk of recurrent VTE and major bleeding in comparison with that on 18 months of placebo. The secondary objectives are: (1) to determine the risk of recurrent VTE after 6 months of warfarin therapy and the presence or the absence of residual lung scan perfusion defect and the persistence or not of elevated D-dimer test; and (2), to determine the impact of extended duration of anticoagulation on the risk of VTE after stopping anticoagulant therapy on a follow-up of 2 years.

Method : French multicenter double blind randomized controlled trial. Inclusion and exclusion criteria and pulmonary diagnostic criteria have been defined. After completing 6 months of oral anticoagulation, a lung scan and D-dimer testing are performed; the investigators and the patients will be unaware of the results of these tests. Then, patients are randomized to receive 18 months of warfarin therapy or 18 months of placebo (the dose of placebo will be adapted according to false computer generated INR). The investigators, the radiologists and the patients are blinded of the treatment allocation. The project will be submitted to national ethical committee and written consent will be obtained from all included patients.

Required number of patients: the expected cumulative frequency of recurrent VTE and major bleeding over 18 months is 4.5% while on warfarin therapy and 16% while on placebo. For a α risk of 5% (to falsely conclude to a true difference) and a β risk of 10% (to falsely conclude to an absence of difference), 178 patients per group should be included. As 5% of patients are expected to be loss, a total of 374 patients is required.

Feasibility: about 50 patients per year are hospitalized in our department of medicine in Brest for an acute episode of idiopathic pulmonary embolism. Four additional centers will participate to the study and have a similar recruitment: HEGP (Pr Meyer, Dr Sanchez), CHU Antoine Béclère (Dr Parent, Pr Simmoneau), CHU Saint Etienne (Pr Mismetti, Pr Décousus), CHU Grenoble (Pr Pison, Pr Carpentier). The study will be coordinated by the Clinical Center of Investigation of Brest Hospital; "true" and "false" INR will be generated by the clinic of anticoagulant of "Ile de France" (Dr Cambus).

Clinical implications: the first consequence of the study is to demonstrate that 6 months of warfarin therapy is inadequate and should be continued for at least 18 additional months after a first episode of idiopathic pulmonary embolism. This study has also the potential to confirm or not the contribution of lung scan and D-dimer testing to appreciate the risk of recurrent VTE after stopping anticoagulant therapy. Lastly, the medical economical impact of such therapeutic management will be evaluated.

DETAILED DESCRIPTION:
Rational: After 3 or 6 months of oral anticoagulation for an episode of acute venous thromboembolism (VTE), the risk of recurrent VTE is high (10 to 15% per year) in comparison with a low risk of recurrence if VTE was provoked by a major transient risk factor such as recent surgery (3% per year) independently of the initial presentation (deep vein thrombosis or pulmonary embolism). After a first episode of idiopathic VTE, 3 months of anticoagulation is associated with a very high risk of recurrence (27% per year); however, the benefit-risk of extended duration of anticoagulation (1 to 2 years) remains uncertain, mainly in relation with an increased risk of anticoagulant related bleeding. Therefore, the last ACCP conference group recommended 6 months of oral anticoagulant therapy after a first episode of idiopathic VTE. However, this recommendation is likely to be inadequate for at least two main reasons: (1) no studies compared 2 years to 6 months of anticoagulation after idiopathic VTE; and (2), if the frequency of recurrent VTE is similar after deep vein thrombosis and pulmonary embolism, however, the case fatality rate of recurrent VTE is higher after pulmonary embolism (12%) than after deep vein thrombosis (5%).

Objective : the main objective is to demonstrate that, after 6 months of oral anticoagulation for a first episode of idiopathic pulmonary embolism, 18 months of warfarin therapy is associated with a lower cumulative risk of recurrent VTE and major bleeding in comparison with that on 18 months of placebo. The secondary objectives are: (1) to determine the risk of recurrent VTE after 6 months of warfarin therapy and the presence or the absence of residual lung scan perfusion defect and the persistence or not of elevated D-dimer test; and (2), to determine the impact of extended duration of anticoagulation on the risk of VTE after stopping anticoagulant therapy on a follow-up of 2 years.

Method : French multicenter double blind randomized controlled trial. Inclusion and exclusion criteria and pulmonary diagnostic criteria have been defined. After completing 6 months of oral anticoagulation, a lung scan and D-dimer testing are performed; the investigators and the patients will be unaware of the results of these tests. Then, patients are randomized to receive 18 months of warfarin therapy or 18 months of placebo (the dose of placebo will be adapted according to false computer generated INR). The investigators, the radiologists and the patients are blinded of the treatment allocation. The project will be submitted to national ethical committee and written consent will be obtained from all included patients.

Required number of patients: the expected cumulative frequency of recurrent VTE and major bleeding over 18 months is 4.5% while on warfarin therapy and 16% while on placebo. For a α risk of 5% (to falsely conclude to a true difference) and a β risk of 10% (to falsely conclude to an absence of difference), 178 patients per group should be included. As 5% of patients are expected to be loss, a total of 374 patients is required.

Feasibility: about 50 patients per year are hospitalized in our department of medicine in Brest for an acute episode of idiopathic pulmonary embolism. Four additional centers will participate to the study and have a similar recruitment: HEGP (Pr Meyer, Dr Sanchez), CHU Antoine Béclère (Dr Parent, Pr Simmoneau), CHU Saint Etienne (Pr Mismetti, Pr Décousus), CHU Grenoble (Pr Pison, Pr Carpentier). The study will be coordinated by the Clinical Center of Investigation of Brest Hospital; "true" and "false" INR will be generated by the clinic of anticoagulant of "Ile de France" (Dr Cambus).

Clinical implications: the first consequence of the study is to demonstrate that 6 months of warfarin therapy is inadequate and should be continued for at least 18 additional months after a first episode of idiopathic pulmonary embolism. This study has also the potential to confirm or not the contribution of lung scan and D-dimer testing to appreciate the risk of recurrent VTE after stopping anticoagulant therapy. Lastly, the medical economical impact of such therapeutic management will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first episode of idiopathic pulmonary embolism who have been treated during 6 months (Plus 30 days or minus 15 days) using Vitamin K antagonist with a INR between 2 and 3.

Exclusion Criteria:

* Age < 18
* warfarin hypersensibility
* unwilling or unable to give written informed consent
* distal or proximal deep vein thrombosis
* Pulmonary embolism which was provoked by a reversible major risk factor
* major thrombophilia (protein C, S or antithrombin deficiency, antiphospholipids antibodies, homozygous factor V Leiden)
* previous documented episode of proximal deep vein thrombosis or pulmonary embolism
* other indication for anticoagulant therapy (e.g.:atrial fibrillation, mechanic valve)
* patient on antithrombotic agent in whom antithrombotic agent should be started again after stopping anticoagulation
* pregnancy
* women without contraception
* planned major surgery in the next 18 months
* ongoing cancer or cured cancer in less than 2 years
* serious bleeding risk (e.g.: gastric ulcer)
* platelet count less than 100 Giga/l
* Life expectancy less than 18 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2007-07; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Symptomatic recurrent venous thromboembolism and serious bleeding | validated standardized objective tests

SECONDARY OUTCOMES:
mortality not due to recurrent venous thromboembolism and bleeding | medical report and death certificates

CONTACTS AND LOCATIONS:
Overall Officials: Francis Couturaud, MD, PhD, Study Chair — Equipe d'Accueil 3878
Locations (1):
- Brest University Hospital, Brest, France

REFERENCES:
- [Derived] Raj L, Presles E, Le Mao R, Robin P, Sanchez O, Pernod G, Bertoletti L, Jego P, Lemarie CA, Leven F, Hoffmann C, Planquette B, Le Roux PY, Slaun PY, Nonent M, Girard P, Lacut K, Melac S, Guegan M, Mismetti P, Laporte S, Meyer G, Leroyer C, Tromeur C, Couturaud F; PADIS-PE Investigators. Evaluation of Venous Thromboembolism Recurrence Scores in an Unprovoked Pulmonary Embolism Population: A Post-hoc Analysis of the PADIS-PE trial. Am J Med. 2020 Aug;133(8):e406-e421. doi: 10.1016/j.amjmed.2020.03.040. Epub 2020 Apr 22. PMID 32333853
- [Derived] Raj L, Robin P, Le Mao R, Presles E, Tromeur C, Sanchez O, Pernod G, Bertoletti L, Jego P, Leven F, Lemarie CA, Martin A, Planquette B, Le Roux PY, Salaun PY, Nonent M, Girard P, Lacut K, Melac S, Mismetti P, Laporte S, Meyer G, Leroyer C, Couturaud F; PADIS-PE Investigators. Predictors for Residual Pulmonary Vascular Obstruction after Unprovoked Pulmonary Embolism: Implications for Clinical Practice-The PADIS-PE Trial. Thromb Haemost. 2019 Sep;119(9):1489-1497. doi: 10.1055/s-0039-1692424. Epub 2019 Jun 23. PMID 31230343
- [Derived] Couturaud F, Sanchez O, Pernod G, Mismetti P, Jego P, Duhamel E, Provost K, dit Sollier CB, Presles E, Castellant P, Parent F, Salaun PY, Bressollette L, Nonent M, Lorillon P, Girard P, Lacut K, Guegan M, Bosson JL, Laporte S, Leroyer C, Decousus H, Meyer G, Mottier D; PADIS-PE Investigators. Six Months vs Extended Oral Anticoagulation After a First Episode of Pulmonary Embolism: The PADIS-PE Randomized Clinical Trial. JAMA. 2015 Jul 7;314(1):31-40. doi: 10.1001/jama.2015.7046. PMID 26151264